CLINICAL TRIAL: NCT03230487
Title: Safety, Tolerability, and Pharmacokinetics of Single (Part 1) and Multiple Rising Oral Doses (Part 2) of BI 1015550 in Healthy Male Subjects
Brief Title: This Study Tests How Healthy Men Tolerate Different Doses of BI1015550. The Study Also Tests How BI 1015550 is Taken up by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1305-0011; 2017-002003-10 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo Single Dose (SD) (Placebo Comparator): Subjects received single dose of placebo tablet matching to BI 1015550 orally with 240 milligram (mL) of water after an overnight fast of at least 10 hours (h) on day 1
  Interventions: Drug: Placebo Single Dose (SD)
- Placebo Multiple Dose (MD) (Placebo Comparator): Subjects received placebo tablet matching to BI 1015550 twice daily (bid) starting on Day 3 orally with 240 milligram (mL) of water after a moderate fat meal. Subjects were treated for 14 days and received a single morning dose on Day 1, followed by 11 day treatment and a single morning dose on Day 14
  Interventions: Drug: Placebo Multiple Dose (MD)
- BI 1015550 36 milligram (mg) Single Dose (SD) (Experimental): Subjects received single dose of BI 1015550 36 mg (6 tablets of 6 mg) orally with 240 milligram (mL) of water after an overnight fast of at least 10 hours (h) on day 1
  Interventions: Drug: BI 1015550 Single Dose (SD)
- BI 1015550 48 milligram (mg) Single Dose (SD) (Experimental): Subjects received single dose of BI 1015550 48 mg (8 tablets of 6 mg) orally with 240 milligram (mL) of water after an overnight fast of at least 10 hours (h) on day 1
  Interventions: Drug: BI 1015550 Single Dose (SD)
- BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) (Experimental): Subjects received BI 1015550 6 mg (1 tablet of 6 mg) twice daily (bid) starting on Day 3 orally with 240 milligram (mL) of water after a moderate fat meal. Subjects were treated for 14 days and received a single morning dose on Day 1, followed by 11 day treatment and a single morning dose on Day 14
  Interventions: Drug: BI 1015550 Multiple Dose (MD)
- BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD) (Experimental): Subjects received BI 1015550 12 mg (2 tablets of 6 mg) twice daily (bid) starting on Day 3 orally with 240 milligram (mL) of water after a moderate fat meal. Subjects were treated for 14 days and received a single morning dose on Day 1, followed by 11 day treatment and a single morning dose on Day 14
  Interventions: Drug: BI 1015550 Multiple Dose (MD)

INTERVENTIONS:
Drug: Placebo Single Dose (SD) — Subjects received single dose of placebo tablet matching to BI 1015550 orally with 240 milligram (mL) of water after an overnight fast of at least 10 hours
  Arms: Placebo Single Dose (SD)
Drug: BI 1015550 Single Dose (SD) — Subjects received single dose of BI 1015550 orally with 240 milligram (mL) of water after an overnight fast of at least 10 hours
  Other Names: Nerandomilast; JASCAYD®
  Arms: BI 1015550 36 milligram (mg) Single Dose (SD); BI 1015550 48 milligram (mg) Single Dose (SD)
Drug: Placebo Multiple Dose (MD) — Subjects received placebo tablet matching to BI 1015550 twice daily (bid) orally with 240 milligram (mL) of water after a moderate fat meal.
  Arms: Placebo Multiple Dose (MD)
Drug: BI 1015550 Multiple Dose (MD) — Subjects received BI 1015550 twice daily (bid) starting on Day 3 orally with 240 milligram (mL) of water after a moderate fat meal.
  Other Names: Nerandomilast; JASCAYD®
  Arms: BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD); BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD)

SUMMARY:
Part 1 (SRD (Single-rising dose)):

The primary objective of this trial part is to investigate the safety and tolerability of BI 1015550 in healthy male subjects following oral administration of single rising doses.

Secondary objectives are the exploration of the pharmacokinetics of BI 1015550 after single dosing.

Part 2 (MRD (Multiple-rising dose)):

In Part 2, the primary objective is to investigate the safety and tolerability of BI 1015550 in healthy male subjects following oral administration of multiple rising doses.

Secondary objectives are the exploration of the pharmacokinetics of BI 1015550 after multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs, 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including vital signs or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 55 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders, including but not limited to mood disorders and any history of suicidality.
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (consumption of more than 20 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until two months after the study completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two months)

In addition, the following trial-specific exclusion criteria apply:

* Positive or missing fecal occult blood (no retest allowed),
* Positive testing for fecal calprotectin (retest allowed)
* Positive testing for hematuria if confirmed by microscopic urine analysis (retest allowed)
* Any lifetime history of suicidal behavior (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior)
* Any suicidal ideation (i.e. type 1-5) on the Columbia Suicidal Severity Rating (C-SSRS) in the past 12 months (i.e.passive/active suicidal thought, active suicidal thought with method, active suicidal thought with intent but without specific plan, or active suicidal thought with plan and intent) (only Part 2)

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Safety, tolerability, and pharmacokinetics of BI 1015550 in healthy male subjects.
  Single rising dose (SRD) part: Partially randomized within dose groups, placebo-controlled, single-blind, parallel-group design; Multiple rising dose (MRD) part: Partially randomized within dose groups, placebo-controlled, double-blind, parallel-group design.
Pre-assignment Details: All subjects were screened for eligibility to participate in the trial. Subjects attended a specialist site which ensured that they (the subjects) met all strictly implemented inclusion/exclusion criteria. Subjects were not to be randomized to trial treatment if any one of the specific entry criteria was violated.
Period: Overall Study
Arm/Group | Placebo Single Dose (SD) | Placebo Multiple Dose (MD) | BI 1015550 36 milligram (mg) Single Dose (SD) | BI 1015550 48 milligram (mg) Single Dose (SD) | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Started | 6 | 8 | 6 | 6 | 8 | 8
Completed | 6 | 8 | 6 | 5 | 8 | 8
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This subject set included all subjects who had received at least 1 dose of trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Single Dose (SD) | Placebo Multiple Dose (MD) | BI 1015550 36 Milligram (mg) Single Dose (SD) | BI 1015550 48 Milligram (mg) Single Dose (SD) | BI 1015550 6 Milligram (mg) Twice Daily Multiple Dose (MD) | BI 1015550 12 Milligram (mg) Twice Daily Multiple Dose (MD) | Total
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 8 | 8 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (7.9) | 33.8 (6.6) | 32.2 (6.6) | 38.2 (7.9) | 35.8 (8.7) | 33.5 (5.3) | 34.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 8 | 6 | 6 | 8 | 8 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was not reported in this trial.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 1 | 0 | 0 | 0 | 2
    White | 6 | 6 | 5 | 6 | 8 | 8 | 39
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug-related Adverse Events (AEs)
Description: Number of subjects with drug-related Adverse Events (AEs).
Time Frame: For SRD: From the administration of study medication until 7 days, up to day 8. For MRD: From the first administration of study medication until 7 days after the last administration of study medication, i.e. up to 21 days after first drug administration.
Population: Treated Set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Single Dose (SD) | Placebo Multiple Dose (MD) | BI 1015550 36 milligram (mg) Single Dose (SD) | BI 1015550 48 milligram (mg) Single Dose (SD) | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Number analyzed (Participants) | 6 | 8 | 6 | 6 | 8 | 8
Participants | 1 | 1 | 2 | 4 | 2 | 4

2. Secondary Outcome: Part 1 (SRD): Area Under the Concentration-time Curve of the BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Part 1 (SRD): Area under the concentration-time curve of the BI 1015550 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Pharmacokinetic samples were taken within 2:00 hours before and 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 34:00, 48:00, 72:00, 96:00, 120:00 hours after drug administration
Population: Pharmacokinetic (PK) parameter set (PKS): This subject set included all subjects of the treated set who provided at least 1 PK parameter that was not excluded because of protocol violations relevant to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/liter (nmol∙h/L)
Arm/Group | BI 1015550 36 milligram (mg) Single Dose (SD) | BI 1015550 48 milligram (mg) Single Dose (SD)
Number analyzed (Participants) | 6 | 5
nanomole*hour/liter (nmol∙h/L) | 5910 (21.2) | 8700 (17.2)

3. Secondary Outcome: Part 1 (SRD): Maximum Measured Concentration of the BI 1015550 in Plasma (Cmax)
Description: Part 1 (SRD): Maximum measured concentration of the BI 1015550 in plasma (Cmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | BI 1015550 36 milligram (mg) Single Dose (SD) | BI 1015550 48 milligram (mg) Single Dose (SD)
Number analyzed (Participants) | 6 | 6
nanomole/liter (nmol/L) | 710 (20.7) | 955 (15.5)

4. Secondary Outcome: Part 2 (MRD) - After the First Dose : Area Under the Concentration-time Curve of the BI 1015550 in Plasma Over a Uniform Dosing Interval Tau After Administration of the First Dose (AUCτ,1)
Description: Part 2 (MRD) - After the first dose : Area under the concentration-time curve of the BI 1015550 in plasma over a uniform dosing interval tau after administration of the first dose (AUCτ,1).
Time Frame: Pharmacokinetic samples were taken within 2:00 hours before and 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 hours after drug administration
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/liter (nmol∙h/L)
Arm/Group | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Number analyzed (Participants) | 8 | 8
nanomole*hour/liter (nmol∙h/L) | 564 (24.8) | 1370 (15.9)

5. Secondary Outcome: Part 2 (MRD) - After the First Dose : Maximum Measured Concentration of the BI 1015550 in Plasma (Cmax)
Description: Part 2 (MRD) - After the first dose : Maximum measured concentration of the BI 1015550 in plasma (Cmax).
Time Frame: Pharmacokinetic samples were taken within 2:00 hours before and 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 34:00, 47:55 hours after drug administration
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Number analyzed (Participants) | 8 | 8
nanomole/liter (nmol/L) | 103 (28.2) | 229 (29.9)

6. Secondary Outcome: Part 2 (MRD) - After the Last Dose: Area Under the Concentration-time Curve of the BI 1015550 in Plasma at Steady State Over a Uniform Dosing Interval Tau (AUCtau,ss)
Description: Part 2 (MRD) - After the last dose: Area under the concentration-time curve of the BI 1015550 in plasma at steady state over a uniform dosing interval tau (AUCtau,ss).
Time Frame: Pharmacokinetic samples were taken within 5 minutes pre-dose and at hours 311:55, 312:15, 312:30, 312:45, 313:00, 313:15, 313:30, 314:00, 315:00, 316:00, 318:00, 320:00, 324:00
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/liter (nmol∙h/L)
Arm/Group | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Number analyzed (Participants) | 8 | 8
nanomole*hour/liter (nmol∙h/L) | 1050 (25.7) | 2300 (15.8)

7. Secondary Outcome: Part 2 (MRD) - After the Last Dose: Maximum Measured Concentration of the BI 1015550 in Plasma at Steady State Over a Uniform Dosing Interval Tau (Cmax,ss)
Description: Part 2 (MRD) - After the last dose: Maximum measured concentration of the BI 1015550 in plasma at steady state over a uniform dosing interval tau (Cmax,ss).
Time Frame: Pharmacokinetic samples were taken within 5 minutes pre-dose and at hours 312:15, 312:30, 312:45, 313:00, 313:15, 313:30, 314:00, 315:00, 316:00, 318:00, 320:00, 324:00, 336:00, 346:00, 360:00, 384:00, 408:00, 432:00, 456:00, 480:00, 504:00
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Number analyzed (Participants) | 8 | 8
nanomole/liter (nmol/L) | 164 (21.3) | 348 (14.1)

8. Secondary Outcome: Part 2 (MRD) - Accumulation Ratio Based on Cmax,ss (RA,Cmax)
Description: Part 2 (MRD) - Accumulation ratio based on Cmax,ss (RA,Cmax). First Dose PK samples were taken within 2:00 hours before and 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 34:00, 47:55 hours after drug administration. Last Dose PK samples were taken within 5 minutes pre-dose and at hours 312:15, 312:30, 312:45, 313:00, 313:15, 313:30, 314:00, 315:00, 316:00, 318:00, 320:00, 324:00, 336:00, 346:00, 360:00, 384:00, 408:00, 432:00, 456:00, 480:00, 504:00.
Time Frame: Up to 504 hours following first drug administration, Please find the time frame in description section.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Number analyzed (Participants) | 8 | 8
Ratio | 1.60 (35.0) | 1.52 (23.6)

9. Secondary Outcome: Part 2 (MRD) - Accumulation Ratio Based on AUC0-tau (RA,AUC)
Description: Part 2 (MRD) - Accumulation ratio based on AUC0-tau (RA,AUC). First Dose PK samples were taken within 2:00 hours before and 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00 hours after drug administration. Last Dose PK samples were taken within 5 minutes pre-dose and at hours 312:15, 312:30, 312:45, 313:00, 313:15, 313:30, 314:00, 315:00, 316:00, 318:00, 320:00, 324:00.
Time Frame: Up to 324 hours following first drug administration, Please find the time frame in description section.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
Number analyzed (Participants) | 8 | 8
Ratio | 1.85 (9.91) | 1.68 (14.8)

ADVERSE EVENTS:
Time Frame: Adverse events: For SRD: From the administration of study medication until 7 days, up to day 8. For MRD: From the first administration of study medication until 7 days after the last administration of study medication, i.e. up to 21 days after first drug administration. All-cause mortality: for SRD, up to 9 days, for MRD, up to 28 days.
Description: Treated set (TS): This subject set included all subjects who had received at least 1 dose of trial medication.
Arm/Group | Placebo Single Dose (SD) | Placebo Multiple Dose (MD) | BI 1015550 36 milligram (mg) Single Dose (SD) | BI 1015550 48 milligram (mg) Single Dose (SD) | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/6 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/6 | 0/6 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 3/8 | 4/6 | 4/6 | 2/8 | 5/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Single Dose (SD) (N=6) | Placebo Multiple Dose (MD) (N=8) | BI 1015550 36 milligram (mg) Single Dose (SD) (N=6) | BI 1015550 48 milligram (mg) Single Dose (SD) (N=6) | BI 1015550 6 milligram (mg) twice daily Multiple Dose (MD) (N=8) | BI 1015550 12 milligram (mg) twice daily Multiple Dose (MD) (N=8)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Occult blood positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 3 | 2 | 3
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/87/NCT03230487/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT03230487/SAP_001.pdf